CLINICAL TRIAL: NCT02181439
Title: Single-center, Controlled, Randomized and Double-blind Study Evaluating the Laser Diode Effect on the Kinetics of Orthodontic Tooth Movement.
Brief Title: Study Evaluating the Laser Diode Effect on the Kinetics of Orthodontic Tooth Movement (Protocol CINELASER)
Acronym: CINELASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC14_0126; 2014-A00471-46 (Other: ANSM)
Record Dates: First submitted 2014-06-27; First posted 2014-07-04 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Class II Canine; Intermaxillary Strength; Elastics II; Multi Fasteners Orthodontic Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right irradiated sector (Other): The low-energy laser (LLLT Low Level Laser Therapy) SIROLaser Advance: laser diode (970nm) is applied twice at day 0 and at M1. For each patient, randomized in this arm, only the right maxillary canine is actually irradiated. Irradiation is performed by scanning an area from the mesial surface of the maxillary canine to the distal surface of the maxillary first molar in the sagittal direction and the cement enamel junction (CEJ) to the bottom of the vestibule in the vertical direction as well in buccally as in Palatine.
  The same procedure will be applied to the left non-irradiated area, the only difference being that the laser will not be activated (placebo, laser inactive). Indeed, only the beam director will be lit and a beep start and end will be heard by the patient. In addition, the practitioner evaluating obtention or not of the class I will not know either which area has been irradiated or not.
  Interventions: Device: (LLLT Low Level Laser Therapy) SiroLaser advance
- Left irradiated sector (Other): The low-energy laser (LLLT Low Level Laser Therapy) SIROLaser Advance: laser diode (970nm) is applied twice at day 0 and at M1. For each patient, randomized in this arm, only the left maxillary canine is actually irradiated. Irradiation is performed by scanning an area from the mesial surface of the maxillary canine to the distal surface of the maxillary first molar in the sagittal direction and the cement enamel junction (CEJ) to the bottom of the vestibule in the vertical direction as well in buccally as in Palatine.
  The same procedure will be applied to the right non-irradiated area, the only difference being that the laser will not be activated (placebo, laser inactive). Indeed, only the beam director will be lit and a beep start and end will be heard by the patient. In addition, the practitioner evaluating obtention or not of the class I will not know either which area has been irradiated or not.
  Interventions: Device: (LLLT Low Level Laser Therapy) SiroLaser advance

INTERVENTIONS:
Device: (LLLT Low Level Laser Therapy) SiroLaser advance — Irradiation scanning distance of the mucosa over an area ranging from the mesial surface of the maxillary canine to the distal surface of the maxillary first molar in the sagittal direction, and the CEJ to the bottom of the vestibule in the vertical direction.

SUMMARY:
It is a single-center, prospective clinical study of a medical device, controlled, randomized, non-stratified, double-blind (neither the patient nor the parents know which area is irradiated / practitioner who performs the measures and evaluates the class I achievement or non also ignores the irradiated area) .

Children included in this clinical trial will be their own control, an area receiving LASER irradiation the other receiving a simulation LASER irradiation (placebo side, inactive laser) .

In the maxilla, it will be segmented using a technique by the introduction of sectional side (portion of elgiloy arch supporting molars, canines and premolars) which serve as a support for Intermaxillary Strength II (or Intermaxillary Elastics II).

The patient should put his own Intermaxillary Elastics II, force adapted to the amount of class II dental, and this 24h/24. The patient should position him/herself these intermaxillary elastics in the first mandibular molar to the maxillary canine ; their action, in case of maximum mandibular anchorage, is to reduce maxillary canine in order to obtain reports of class I. In the mandible, a maximum anchor will be realized. Maximum molar anchor is to place the roots of mandibular molars in the vestibular cortex in order to anchor them there. This allows the lower canines, premolars and maxillary molars under the action of FIM without causing mutual advancement of the mandibular arch.

This procedure does not differ from the usual treatment. The application of laser diode appears, by biomodulatrice action, to show promising results on accelerating the kinetics of tooth movement during orthodontic treatment. The main hypothesis of the research is an increase in the rate of correction of Class II irradiated side, i.e. a 1-month shortest delay in obtaining the class I for irradiated areas vs. non irradiated ones.

The main objective of this study is to evaluate the effect of the application of low energy laser (LLLT) on the time required to obtain a Class I canine on patients undergoing FIM II (Class II elastics)

ELIGIBILITY:
Pre-inclusion criteria:

Written consent of parental authority, ie if any of the two parents, will be required, but the apparent unwillingness of the child shall prevail if any.

No exclusion period is required if the child has already attended another biomedical research.

Inclusion criteria:

* With a Class II canine complete or partial, bilateral and symmetrical
* In permanent dentition (no deciduous teeth in the arch)
* Requiring the use of intermaxillary strength (FIM) II correction dental class II during a multi fasteners orthodontic treatment
* Leveling done beforehand*
* Anchor of the mandible is maximum

  * The same technique employed should be segmented in the maxilla, in all patients (lateral sectional canine to molar).

Exclusion Criteria:

Patient :

* having a mental deficiency or child who can not read or write (difficulties in completing the questionnaire )
* with lack of cooperation (withdrawal, refuse to wear FIM II)
* who missed at least 3 consecutive appointments according to the medical record ,
* with orofacial malignant tumor
* having unbalanced chronic diseases or patient receiving treatment that can interfere with orthodontic treatment or with pain assessment (antibiotics, analgesics, treatment of bone and mineral metabolism, diabetes, hormonal treatments excluding contraceptives)
* with a Class II dental unilateral and asymmetric
* with a dental anomaly from shape and / or structure related to the following teeth: maxillary canines and first molars causing an increased risk of detachment brackets
* with anomalies of number : agenesis of permanent teeth
* with a mixed dentition
* refusing to give consent or with one or two parents refusing to give their consent (for minor patients)
* participating in another biomedical research
* pregnant

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Delays in obtaining Class I canine right and left | 6 months
  For each sector, obtaining or not the class I will be assessed each month up to 6 months. The difference of delay in obtaining Class I between sectors will be calculated for each patient. For this reason, the primary outcome assessment will be done after 6 months of follow-up + 18 months of inclusion period, i.e. 24 months after starting inclusions.The comparison will be made from a student test on the difference in time required to obtain Class I between sectors.
  If class I is obtained on each sector (right and left) prior to the 6-month FUp, the corresponding visit is considered as the last one for the patient within the study.

SECONDARY OUTCOMES:
Total distance covered by the maxillary canine (mm) until the Class I canine | 6 months
  The total distance until the class I will be collected for each sector and will be compared using a student test.
Intensity pain jaw | 6 months
  Intensity pain jaw while wearing FIM II = quantitative pain assessment in the maxilla via EVA, by right and left during the first 3 days of FIM II port via a patient diary Jaw pain felt in each sector will be collected over 3 days. Comparison to be made each time from a student test on the difference in jaw pain felt across sectors.
speed in obtaining Class I canine right and left | 6 months
  total distance until the class I/ Delay in obtaining Class I

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NANTES - Service d'odontologie restauratrice et chirurgicale, UIC odontologie, Nantes, France

REFERENCES:
- [Derived] Perignon B, Bandiaky ON, Fromont-Colson C, Renaudin S, Pere M, Badran Z, Cuny-Houchmand M, Soueidan A. Effect of 970 nm low-level laser therapy on orthodontic tooth movement during Class II intermaxillary elastics treatment: a RCT. Sci Rep. 2021 Dec 1;11(1):23226. doi: 10.1038/s41598-021-02610-7. PMID 34853360